CLINICAL TRIAL: NCT03057197
Title: The Influence of Needle-insertion Depth on Successful Epidurogram and Clinical Outcome in Caudal Epidural Injections: A Randomized Clinical Trial
Brief Title: The Influence of Needle-insertion Depth on Successful Epidurogram and Clinical Outcome in Caudal Epidural Injections
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The results of the interim analysis showed significant results.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 4-2016-1030
Record Dates: First submitted 2017-02-15; First posted 2017-02-17 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Lumbosacral Radicular Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (No Intervention): Conventional method group (n=85): caudal injection after advancement of the needle into the sacral canal. Ultrasound is used to achieve accurate needle placement and we will check intravascular injection using digital subtraction angiography.
- Group B (Experimental): New method group (n=85): same as conventional method group except caudal injection right after penetrating the sacrococcygeal ligament.
  Interventions: Procedure: new caudal injection technique

INTERVENTIONS:
Procedure: new caudal injection technique — new caudal injection technique is applied to the Group B, which is that the needle only penetrates the sacrococcygeal ligament without being inserted into the sacral canal
  Arms: Group B

SUMMARY:
Caudal epidural injections have been commonly performed in patients with low back pain and radiculopathy. Conventional caudal epidural injections, which the needle is advanced into the sacral canal, present a potential risk of penetration of the epidural venous plexus or dura. The investigators hypothesized that a new caudal injection technique, which the needle only penetrates the sacrococcygeal ligament without being inserted into the sacral canal, might represent a safe alternative, with a lower incidence of intravascular injections and patient's discomfort during the procedure than the conventional technique. The study is designed to investigate the influence of the depth of the inserted needle on successful epidurogram and clinical outcome in caudal epidural injections under the ultrasound and digital subtraction angiography.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (20-80 years of age) who were scheduled to receive caudal epidural injection for lumbosacral radicular pain at our pain management clinic

Exclusion Criteria:

* pregnancy
* coagulopathy
* systemic infection
* any active infection at the injection site
* history of allergy to contrast media, local anesthetics, corticosteroid
* patients unable to communicate or patients with cognitive dysfunction

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2018-04-23 (Actual); Study Completion 2018-04-23 (Actual)

PRIMARY OUTCOMES:
the incidence of intravascular injection | 5 seconds after injection of contrast media via block needle.
  the incidence of intravascular injection in the conventional method group and the new method group during the caudal epidural injections.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University College of Medicine, Department of internal Medicine, Division of Endocrinology, Severance Hospital, Diabetes Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No